CLINICAL TRIAL: NCT02524730
Title: Scorpio NRG Prospective, Open-label, Post-market International Multicentre Outcome Study
Brief Title: Scorpio NRG (eNeRGize) Cruciate Retaining (CR) Post-market International Outcome Study
Acronym: Scorpio NRG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SLCRG-001-2007 / K-S-002
Record Dates: First submitted 2015-06-11; First posted 2015-08-17 (Estimated); Results first posted 2021-06-14 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Scorpio NRG CR Total Knee System (Other): Primary total knee replacement
  Interventions: Device: Primary total knee replacement (Scorpio NRG CR Total Knee System)

INTERVENTIONS:
Device: Primary total knee replacement (Scorpio NRG CR Total Knee System) — Scorpio NRG CR Total Knee System

SUMMARY:
The purpose of this study is to collect basic function, radiographic and patient satisfaction data for observation and analysis.

DETAILED DESCRIPTION:
Evaluation of the effect of the component design on functional performance by comparing postoperative Knee Society Scores (KSS) with preoperative.

Evaluate post-operative radiographic findings. Evaluate the effect of component design on patient activity by comparing postoperative Lower Extremity Activity Scale (LEAS) with preoperative.

Evaluate patient satisfaction using Short-Form-36 Health Survey (SF-36). Evaluate quality of life using Knee Injury and Osteoarthritis Outcome Score (KOOS) and EuroQuol-5 dimension patient questionaire (EQ-5D).

ELIGIBILITY:
Inclusion Criteria:

1. Patient is able to understand the meaning of the study and is willing to sign the Ethic Commission approved, study specific Informed Patient Consent Form.
2. The subject is a male or non-pregnant female between 40 and 75 years of age.
3. The subject requires a primary total knee replacement.
4. Patients with osteoarthritis or posttraumatic arthritis (no rheumatoid arthritis)
5. The subject has intact collateral ligaments.
6. The subject is willing and able to comply with postoperative scheduled clinical and radiographic evaluations and rehabilitation.
7. The subject is capable of understanding the patient scores in the national language.

Exclusion Criteria:

1. The subject is morbidly obese, defined as Body Mass Index (BMI) of > 40.
2. The subject has a history of total or unicompartmental reconstruction of the affected joint.
3. The subject will be operated bilaterally.
4. Patients who had a Total Hip Arthroplasty (THA) on contralateral and/or ipsilateral side within the last year that is considered to have an unsatisfactory outcome (Patients with contralateral and/or ipsilateral THA > 1 year ago with good outcome can be included in the study).
5. Patients who had a Total Knee Arthroplasty (TKA) on contralateral side within the last 6 months that is considered to have an unsatisfactory outcome. (Patients with contralateral TKA > 6 months ago with good outcome can be included in the study).
6. Patients who will need lower limb joint replacement for another joint within one year.
7. The subject has had a high tibial osteotomy or femoral osteotomy.
8. The subject has a neuromuscular or neurosensory deficiency, which would limit the ability to assess the performance of the device.
9. The subject has a systemic or metabolic disorder leading to progressive bone deterioration.
10. The subject is immunologically suppressed or receiving steroids in excess of normal physiological requirements.
11. The subject's bone stock in compromised by disease or infection which cannot provide adequate support and/or fixation to the prosthesis.
12. The subject has had a knee fusion to the affected joint.
13. The subject has an active or suspected latent infection in or about the knee joint.
14. Proven or suspected hypersensitivity to one or more than one of the device materials (see Appendix 10 table of chemical composition).
15. Female patients planning a pregnancy during the course of the study.
16. The subject is a prisoner.
17. severe deformities: varus/valgus deformity >10° (mech. axis), bowed femur > 20 degree, flexion contracture >10°

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2009-05-18 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Krismer, Prof., Principal Investigator — Medical University Innsbruck
Locations (5):
- Medical University Hospital Innsbruck, Innsbruck, Tyrol, Austria
- Knappschaftskrankenhaus Dortmund, Dortmund, North Rhine-Westphalia, Germany
- Netherlands (2):
  - Orthopaedische Maatschap Leeuwarden, Leeuwarden, Provincie Friesland
  - St. Antonius Ziekenhuis, Nieuwegein, Utrecht
- Royal Devon and Exeter NHS Foundation Trust, Exeter, Devon, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 205 participants who agreed to participate in the study following completion of the informed consent process were enrolled into the study
Period: Overall Study
Arm/Group | Scorpio NRG CR Total Knee System
Started | 205
Completed | 159
Not Completed | 46
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 18
Not completed — Death | 10
Not completed — Adverse Event | 8
Not completed — Protocol Violation | 1
Not completed — Subjects received Scorpio NRG PS (Posterior Stabilizing) | 4

BASELINE CHARACTERISTICS:
Arm/Group | Scorpio NRG CR Total Knee System
Number analyzed (Participants) | 205
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.53 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Gender information permanently missing in one case.
  Participants
    number analyzed (Participants) | 204
    Female | 132
    Male | 72
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Europe | 205
Indication [Number; unit: participants] — Population: Indication information permanently missing in one case.
  participants
    Osteoarthritis: number analyzed (Participants) | 204
    Osteoarthritis | 200
    Post-traumatic Arthritis: number analyzed (Participants) | 204
    Post-traumatic Arthritis | 4

OUTCOME MEASURES:

1. Primary Outcome: Survival Rate
Description: Assess survival (absence of revision) at 7 year follow-up
Time Frame: 7 year follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Scorpio NRG CR Total Knee System
Number analyzed (Participants) | 197
Participants
  Femoral Component Revision | 2
  Inlay Revision | 1
  Tibial Tray Revision | 1
  Total Knee Arthroplasty Revision | 4
  No Revision | 189

2. Secondary Outcome: Investigation of Clinical Performance and Patient Outcome With the Knee Society Score (KSS)
Description: The Knee Society Clinical Rating System is comprised of two distinct sub-scores: one for pain, range of motion (ROM) and joint stability, and one for functional parameters. Sub-scores range from a potential minimum score of 0 to a maximum score of 100 points. Although the specific scores are not distinguished as "excellent," "good," "fair," or "poor," a higher value represents a better outcome.
Time Frame: Pre-operative, 3 months, 1, 3, 5 and optional 7 years
Population: Numbers analyzed represent evaluable cases
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Scorpio NRG CR Total Knee System
Number analyzed (Participants) | 204
units on a scale
  Pre-operative pain motion score: number analyzed (Participants) | 202
  Pre-operative pain motion score | 57.84 (13.34)
  Pain motion score at 3 months: number analyzed (Participants) | 195
  Pain motion score at 3 months | 78.71 (12.36)
  Pain motion score at 1 year: number analyzed (Participants) | 187
  Pain motion score at 1 year | 83.27 (10.15)
  Pain motion score at 3 years: number analyzed (Participants) | 177
  Pain motion score at 3 years | 83.85 (11.42)
  Pain motion score at 5 years: number analyzed (Participants) | 164
  Pain motion score at 5 years | 84.73 (11.57)
  Pain motion score at 7 years: number analyzed (Participants) | 142
  Pain motion score at 7 years | 84.20 (10.33)
  Pre-operative function score | 61.54 (17.78)
  Function score at 3 months: number analyzed (Participants) | 195
  Function score at 3 months | 78.05 (16.95)
  Function score at 1 year: number analyzed (Participants) | 187
  Function score at 1 year | 87.99 (15.68)
  Function score at 3 years: number analyzed (Participants) | 180
  Function score at 3 years | 85.00 (19.34)
  Function score at 5 years: number analyzed (Participants) | 164
  Function score at 5 years | 83.75 (19.75)
  Function score at 7 years: number analyzed (Participants) | 144
  Function score at 7 years | 83.51 (21.43)

3. Secondary Outcome: Investigation of Clinical Performance and Patient Outcome With the Lower Extremity Activity Scale (LEAS) Patient Questionnaire
Description: The LEAS is completed by the participant to assess activity level. Activity levels were ordered in terms of intensity from 1 to 18, with 18 indicating the highest activity level.
Time Frame: Pre-operative, 3 months,1, 3, 5 and optional 7 years
Population: Numbers analyzed represent evaluable cases.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Scorpio NRG CR Total Knee System
Number analyzed (Participants) | 205
units on a scale
  pre-operative activity level: number analyzed (Participants) | 204
  pre-operative activity level | 8.61 (2.51)
  Activity level at 3 months: number analyzed (Participants) | 194
  Activity level at 3 months | 9.43 (2.81)
  Activity level at 1 year: number analyzed (Participants) | 186
  Activity level at 1 year | 11.11 (3.06)
  Activity level at 3 years: number analyzed (Participants) | 176
  Activity level at 3 years | 10.68 (3.00)
  Activity level at 5 years: number analyzed (Participants) | 154
  Activity level at 5 years | 10.38 (3.09)
  Activity level at 7 years: number analyzed (Participants) | 133
  Activity level at 7 years | 10.75 (3.20)

4. Secondary Outcome: Investigation of Clinical Performance and Patient Outcome With the Short Form - 36 Health Survey (SF-36)
Description: The SF-36 is a 36-item patient completed questionnaire to measure general health and well-being. It includes physical and mental status component sub scores (physical function, physical role functioning, body pain, general health, vitality, social functioning, emotional role, mental health); each ranging from 0-100. Low values represent a poor health state and high values represent a good health state.
Time Frame: Pre-operative, 3 months,1, 3, 5 and optional 7 years
Population: Numbers analyzed represent evaluable cases.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Scorpio NRG CR Total Knee System
Number analyzed (Participants) | 205
units on a scale
  Pre-operative physical function: number analyzed (Participants) | 193
  Pre-operative physical function | 30.62 (7.91)
  Physical function at 3 months: number analyzed (Participants) | 186
  Physical function at 3 months | 40.2 (8.86)
  Physical function at 1 year: number analyzed (Participants) | 180
  Physical function at 1 year | 44.67 (8.6)
  Physical function at 3 years: number analyzed (Participants) | 169
  Physical function at 3 years | 43.97 (9.8)
  Physical function at 5 years: number analyzed (Participants) | 161
  Physical function at 5 years | 42.41 (10.8)
  Physical function at 7 years: number analyzed (Participants) | 132
  Physical function at 7 years | 43.07 (10.71)
  Pre-operative physical role functioning: number analyzed (Participants) | 198
  Pre-operative physical role functioning | 34.48 (9.19)
  Physical role functioning at 3 months: number analyzed (Participants) | 193
  Physical role functioning at 3 months | 39.04 (9.34)
  Physical role functioning at 1 year: number analyzed (Participants) | 186
  Physical role functioning at 1 year | 45.11 (9.77)
  Physical role functioning at 3 years: number analyzed (Participants) | 177
  Physical role functioning at 3 years | 44.0 (9.77)
  Physical role functioning at 5 years: number analyzed (Participants) | 165
  Physical role functioning at 5 years | 43.26 (10.75)
  Physical role functioning at 7 years: number analyzed (Participants) | 141
  Physical role functioning at 7 years | 43.65 (10.56)
  Pre-operative body pain: number analyzed (Participants) | 193
  Pre-operative body pain | 42.24 (3.23)
  Body pain at 3 months: number analyzed (Participants) | 190
  Body pain at 3 months | 40.69 (3.52)
  Body pain at 1 year: number analyzed (Participants) | 185
  Body pain at 1 year | 39.72 (3.28)
  Body pain at 3 years: number analyzed (Participants) | 177
  Body pain at 3 years | 39.47 (3.17)
  Body pain at 5 years: number analyzed (Participants) | 165
  Body pain at 5 years | 39.48 (3.74)
  Body pain at 7 years: number analyzed (Participants) | 142
  Body pain at 7 years | 39.35 (3.3)
  Pre-operative general health: number analyzed (Participants) | 198
  Pre-operative general health | 49.2 (8.15)
  General health at 3 months: number analyzed (Participants) | 190
  General health at 3 months | 51.48 (7.57)
  General health at 1 year: number analyzed (Participants) | 186
  General health at 1 year | 51.6 (8.28)
  General health at 3 years: number analyzed (Participants) | 177
  General health at 3 years | 49.9 (8.38)
  General health at 5 years: number analyzed (Participants) | 165
  General health at 5 years | 48.95 (9.02)
  General health at 7 years: number analyzed (Participants) | 140
  General health at 7 years | 48.11 (8.82)
  Pre-operative vitality: number analyzed (Participants) | 200
  Pre-operative vitality | 49.94 (8.61)
  Vitality at 3 months: number analyzed (Participants) | 192
  Vitality at 3 months | 52.73 (8.93)
  Vitality at 1 year: number analyzed (Participants) | 183
  Vitality at 1 year | 55.71 (9.4)
  Vitality at 3 years: number analyzed (Participants) | 177
  Vitality at 3 years | 54.61 (9.46)
  Vitality at 5 years: number analyzed (Participants) | 165
  Vitality at 5 years | 54.42 (8.56)
  Vitality at 7 years: number analyzed (Participants) | 140
  Vitality at 7 years | 54.52 (9.38)
  Pre-operative social functioning: number analyzed (Participants) | 201
  Pre-operative social functioning | 44.67 (10.12)
  Social functioning at 3 months: number analyzed (Participants) | 191
  Social functioning at 3 months | 49.17 (8.91)
  Social functioning at 1 year: number analyzed (Participants) | 185
  Social functioning at 1 year | 51.16 (8.54)
  Social functioning at 3 years: number analyzed (Participants) | 178
  Social functioning at 3 years | 51.27 (8.26)
  Social functioning at 5 years: number analyzed (Participants) | 165
  Social functioning at 5 years | 50.83 (7.96)
  Social functioning at 7 years: number analyzed (Participants) | 142
  Social functioning at 7 years | 49.97 (8.98)
  Pre-operative emotional role: number analyzed (Participants) | 198
  Pre-operative emotional role | 43.41 (12.92)
  Emotional role at 3 months: number analyzed (Participants) | 193
  Emotional role at 3 months | 46.65 (11.65)
  Emotional role at 1 year: number analyzed (Participants) | 185
  Emotional role at 1 year | 47.81 (11.10)
  Emotional role at 3 years: number analyzed (Participants) | 177
  Emotional role at 3 years | 46.83 (10.81)
  Emotional role at 5 years: number analyzed (Participants) | 165
  Emotional role at 5 years | 47.47 (11.4)
  Emotional role at 7 years: number analyzed (Participants) | 142
  Emotional role at 7 years | 46.0 (11.78)
  Pre-operative mental health: number analyzed (Participants) | 200
  Pre-operative mental health | 50.23 (9.4)
  Mental health at 3 months: number analyzed (Participants) | 191
  Mental health at 3 months | 52.6 (9.86)
  Mental health at 1 year: number analyzed (Participants) | 184
  Mental health at 1 year | 53.39 (9.96)
  Mental health at 3 years: number analyzed (Participants) | 175
  Mental health at 3 years | 53.06 (8.80)
  Mental health at 5 years: number analyzed (Participants) | 165
  Mental health at 5 years | 53.52 (8.63)
  Mental health at 7 years: number analyzed (Participants) | 140
  Mental health at 7 years | 52.5 (9.36)

5. Secondary Outcome: Investigation of Clinical Performance and Patient Outcome With the Knee Injury and Osteoarthritis Outcome Score (KOOS) Patient Questionnaire.
Description: KOOS consists of 5 subscales: Pain, other symptoms, function in daily living , function in sport and recreation and knee related quality of life (QOL). The previous week is the time period considered when answering the questions. Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms).
Time Frame: Pre-operative,1, 5 and optional 7 years
Population: Numbers analyzed represent evaluable cases. The KOOS was collected pre-operatively and at 1, 5 and 7 years only.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Scorpio NRG CR Total Knee System
Number analyzed (Participants) | 202
units on a scale
  Symptoms pre-operative | 49.91 (18.55)
  Symptoms at 1 year: number analyzed (Participants) | 184
  Symptoms at 1 year | 79.58 (15.73)
  Symptoms at 5 years: number analyzed (Participants) | 165
  Symptoms at 5 years | 83.38 (16.1)
  Symptoms at 7 years: number analyzed (Participants) | 144
  Symptoms at 7 years | 85.83 (15.46)
  Pain pre-operative: number analyzed (Participants) | 201
  Pain pre-operative | 41.28 (17.82)
  Pain at 1 year: number analyzed (Participants) | 184
  Pain at 1 year | 82.9 (19.14)
  Pain at 5 years: number analyzed (Participants) | 165
  Pain at 5 years | 84.36 (19.38)
  Pain at 7 years: number analyzed (Participants) | 144
  Pain at 7 years | 86.99 (17.74)
  Function, sports and recreation activities pre-operative | 14.15 (16.26)
  Function, sports and recreation activities at 1 year: number analyzed (Participants) | 177
  Function, sports and recreation activities at 1 year | 47.89 (29.08)
  Function, sports and recreation activities at 5 years: number analyzed (Participants) | 164
  Function, sports and recreation activities at 5 years | 48.71 (31.05)
  Function, sports and recreation activities at 7 years: number analyzed (Participants) | 140
  Function, sports and recreation activities at 7 years | 52.79 (33.45)
  Quality of life (QoL) pre-operative | 24.36 (14.86)
  QoL at 1 year: number analyzed (Participants) | 182
  QoL at 1 year | 66.19 (24.11)
  QoL at 5 years: number analyzed (Participants) | 165
  QoL at 5 years | 66.78 (23.41)
  QoL at 7 years: number analyzed (Participants) | 144
  QoL at 7 years | 65.54 (21.81)
  Function, daily living pre-operative: number analyzed (Participants) | 201
  Function, daily living pre-operative | 46.59 (18.2)
  Function, daily living at 1 year: number analyzed (Participants) | 183
  Function, daily living at 1 year | 82.7 (17.35)
  Function, daily living at 5 years: number analyzed (Participants) | 165
  Function, daily living at 5 years | 83.47 (18.46)
  Function, daily living at 7 years: number analyzed (Participants) | 144
  Function, daily living at 7 years | 84.24 (19.23)

6. Secondary Outcome: Investigation of Clinical Performance and Patient Outcome With the EuroQuol-5 Dimension Health Questionnaire (EQ-5D).
Description: The EuroQol-5 Dimension (EQ-5D) is a subject-completed questionnaire designed to assess subject health state values. The EQ-5D consists of 2 areas; EQ-5D descriptive system and the visual analogue scale (VAS). The EQ-5D descriptive system comprises the following five dimensions: mobility self care, usual activities, pain/comfort and anxiety/depression. Each dimension has 3 levels indicating no problems, some problems or extreme problems. The index values on a scale between -1 (low) and 1 (high) are showing the average health status according to the 5 dimensions: A low score shows worse health and a high score shows better health.
  With the EQ VAS the respondents can report their perceived health status with a grade ranging from 0 (the worst possible health status) to 100 (the best possible health status).
Time Frame: Pre-operative, 3 months,1, 3, 5 and optional 7 years
Population: Numbers analyzed represent evaluable cases.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Scorpio NRG CR Total Knee System
Number analyzed (Participants) | 203
units on a scale
  Pre-operative visual analogue scale (VAS): number analyzed (Participants) | 200
  Pre-operative visual analogue scale (VAS) | 70.97 (16.75)
  VAS at 3 months: number analyzed (Participants) | 190
  VAS at 3 months | 76.96 (13.92)
  VAS at 1 year: number analyzed (Participants) | 187
  VAS at 1 year | 77.41 (14.40)
  VAS at 3 years: number analyzed (Participants) | 177
  VAS at 3 years | 75.09 (14.11)
  VAS at 5 years: number analyzed (Participants) | 165
  VAS at 5 years | 76.84 (13.23)
  VAS at 7 years: number analyzed (Participants) | 144
  VAS at 7 years | 77.03 (14.77)
  Pre-operative descriptive EQ-5D | 0.55 (0.26)
  Descriptive EQ-5D at 3 months: number analyzed (Participants) | 191
  Descriptive EQ-5D at 3 months | 0.77 (0.17)
  Descriptive EQ-5D at 1 year: number analyzed (Participants) | 185
  Descriptive EQ-5D at 1 year | 0.84 (0.17)
  Descriptive EQ-5D at 3 years: number analyzed (Participants) | 175
  Descriptive EQ-5D at 3 years | 0.83 (0.19)
  Descriptive EQ-5D at 5 years: number analyzed (Participants) | 163
  Descriptive EQ-5D at 5 years | 0.82 (0.20)
  Descriptive EQ-5D at 7 years: number analyzed (Participants) | 144
  Descriptive EQ-5D at 7 years | 0.83 (0.19)

ADVERSE EVENTS:
Time Frame: Recording of Adverse Events ongoing from when the subject has signed the informed consent up to 5 years follow-up or optional 7 years follow-up.
Arm/Group | Scorpio NRG CR Total Knee System
All-Cause Mortality (participants affected / at risk) | 10/205
Serious Adverse Events (participants affected / at risk) | 88/205
Other Adverse Events (participants affected / at risk) | 15/205
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Scorpio NRG CR Total Knee System (N=205)
Quadriceps tendon rupture (Musculoskeletal and connective tissue disorders) | 1 (2)
Inlay wear (Musculoskeletal and connective tissue disorders) | 1 (1)
Instability (Musculoskeletal and connective tissue disorders) | 2 (2)
Aseptic loosening (Musculoskeletal and connective tissue disorders) | 2 (2)
Post cruciate ligament rupture (Musculoskeletal and connective tissue disorders) | 2 (2)
Great toe surgery (Musculoskeletal and connective tissue disorders) | 3 (4)
Retropatellar arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 5 (6)
Shoulder tendon rupture (Musculoskeletal and connective tissue disorders) | 1 (1)
Carpal tunnel syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Hemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Elbow fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Per-trochanteric fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Knee pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Ankle arthrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Patella subluxation (Musculoskeletal and connective tissue disorders) | 1 (1)
Adhesion (Musculoskeletal and connective tissue disorders) | 1 (1)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 17 (18)
Myocard infarction (Cardiac disorders) | 7 (7)
Heart valve disease (Cardiac disorders) | 2 (2)
Cardiovascular collapse (Cardiac disorders) | 2 (2)
Coronary artery disease (Cardiac disorders) | 3 (3)
Cehst pain (Cardiac disorders) | 1 (1)
Heart failure and dyspnea (Cardiac disorders) | 1 (1)
Diverticulitis (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Suicide (General disorders) | 1 (1)
General health issues (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Hepatitis E (Hepatobiliary disorders) | 1 (1)
Polyarteritis nodosa (Immune system disorders) | 1 (1)
Pneumonia infections (Infections and infestations) | 4 (4)
Deep joint infection (Infections and infestations) | 1 (1)
pre-patellar bursitis (Infections and infestations) | 1 (1)
head/spinal cord trauma (Injury, poisoning and procedural complications) | 2 (2)
Wound dehiscence/hematoma (Injury, poisoning and procedural complications) | 2 (2)
Death unknown cause (General disorders) | 2 (2)
Dementia (Nervous system disorders) | 1 (1)
Fraxiparine allergy (Product Issues) | 1 (1)
Kidney stone (Renal and urinary disorders) | 1 (1)
COPD (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Necrotic wound (Skin and subcutaneous tissue disorders) | 1 (1) — not operative site related
Posterior intervaginal plasty (Surgical and medical procedures) | 1 (1)
Pulmonary embolism (Vascular disorders) | 1 (1)
Stroke (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Scorpio NRG CR Total Knee System (N=205)
Knee pain (Musculoskeletal and connective tissue disorders) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-09): https://cdn.clinicaltrials.gov/large-docs/30/NCT02524730/Prot_SAP_000.pdf